CLINICAL TRIAL: NCT02569112
Title: Prospective Internally Controlled Blind Reviewed Clinical Evaluation of Cryolipolysis Combined With MP2 Technology for Enhanced Subject Results in Circumferential Fat Reduction and Skin Laxity of the Flanks
Brief Title: Evaluation of CoolSculpt Combining Venus Legacy Technology for Enhanced Results in Fat Reduction & Laxity of the Flanks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CS0915
Record Dates: First submitted 2015-08-24; First posted 2015-10-06 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2017-12

CONDITIONS: Adipose Tissue

STUDY DESIGN:
Intervention Model Description: All participants to receive cryolipolysis treatment on one side of their body and cryolipolysis plus multipolar radiofrequency with varipulse technology treatment on the other side of their body.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both investigator and independent reviewer to determine which side of the body the multi-polar radiofrequency, pulsed-electromagnetic fields and vacuum therapy was applied.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cryolipolysis (Active Comparator): Each patient is their own control and one side will have only a cryolipolysis treatment while the other side will have a cryolipolysis treatment plus multipolar radiofrequency and varipulse treatment.
  Interventions: Device: cryolipolysis
- cryolipolysis, multipolar RF, varipulse (Experimental): Each patient is their own control and one side will have only a cryolipolysis treatment while the other side will have a cryolipolysis treatment plus multipolar radiofrequency and varipulse treatment.
  Interventions: Device: multipolar RF, varipulse; Device: cryolipolysis

INTERVENTIONS:
Device: multipolar RF, varipulse — Multi-polar Radio frequency (RF) technology combining pulsed electro magnetic fields (PEMF) and mild suction stimulation (varipulse).
  Other Names: Venus Legacy
  Arms: cryolipolysis, multipolar RF, varipulse
Device: cryolipolysis — Cryolipolysis technology uses the sensitivity of fat cells to cold injury, causing them to freeze and undergo cellular apoptosis.
  Other Names: CoolSculpt

SUMMARY:
The purpose of this study is to evaluate the effect on the subject outcome using the combination of the Zeltiq Cryolipolysis device and the Venus Concept multipolar radiofrequency device with varipulse technology for the enhanced non-surgical treatment of skin laxity in the flank area.

DETAILED DESCRIPTION:
Commercially available as the Zeltiq CoolSculpting system, cryolipolysis is FDA cleared for use in the United States for an indication of fat layer reduction in the flanks, thighs, and abdomen through cold-assisted lipolysis. CoolSculpting has been clinically proven to non-surgically reduce subcutaneous fat bulges, allowing patients to achieve noticeable and measurable aesthetic results without the pain, expense, downtime, and risks associated with existing invasive and minimally-invasive procedures. The Zeltiq CoolSculpting System is a non-invasive device designed to cool subcutaneous fat without affecting adjacent or underlying structures.

The RF device to be used in this study is a FDA cleared device used for aesthetic non-surgical skin tightening procedures including wrinkles, skin rhytides and cellulite in the face and body. The Venus Legacy utilizes a multi-polar radiofrequency system to deliver homogenous heating to multiple tissue depths. The Venus Legacy device also utilizes pulsed magnetic field technology as well as pulsed negative pressure technology.

The flanks of Ten (10) healthy adults (male and female), 21 to 50 years of age, who desire a reduction in focal fat of the flanks will be recruited from the investigator's subject populations. Informed Consent will be obtained from each subject during a screening visit.

The photos will be taken prior to the treatment series, one week post treatment series, at 3 and 6 months post treatment series for the evaluation of two blinded reviewers as well as for the investigator to assess.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.
* Subjects who have pre-scheduled a body contouring procedure.
* Subjects have clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
* Subjects have not had weight change exceeding 10 pounds in the preceding month.
* Subjects agree to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.

Exclusion Criteria:

* Subjects with active localized or systemic infections.
* Immuno-compromised subjects.
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* In the opinion of the trained clinician, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Subjects with a history of radiation therapy to the treatment area.
* Subjects with any skin pathology or condition that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments.
* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject has a history of hernia in the areas to be treated.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Few, MD, Principal Investigator — Few Institute
Locations (1):
- Few Institute, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten subjects between the ages of 21 and 50 years of age, requesting a reduction in focal fat of the flanks were recruited from a single outpatient clinic.
Pre-assignment Details: Subjects received one session of cryolipolysis treatment on both sides of their body before one side of their body was treated with multipolar radiofrequency plus varipulse technology. Each subject acted as their own control.
Units Other Than Participants: flanks
Groups:
- Cyrolipolysis: Each side of the subject received a cryolipolysis treatment.
- Cryolipolysis, Multipolar RF With Varipulse Technology: One side of the body received cryolipolysis plus multipolar radiofrequency with varipulse technology
Period: Overall Study
Arm/Group | Cyrolipolysis | Cryolipolysis, Multipolar RF With Varipulse Technology
Started | 10; 20 flanks | 10; 10 flanks
Completed (Each subject received a single cryolipolysis treatment on both sides of their body.) | 10; 20 flanks | 10; 10 flanks (Each subject received multipolar RF with varipulse technology to only one side of their body.)
Not Completed | 0; 0 flanks | 0; 0 flanks

BASELINE CHARACTERISTICS:
Population: Each subject received a cryolipolysis treatment to both sides of body. One side of the flank will then receive multipolar RF and PEMF with Varipulse technology and the other side will not.
Units Other Than Participants: flanks
Groups:
- Cryolipolysis Treatment & Cryolipolysis With Legacy: Each patient is their own control. Both flanks will be treated with cryolypolysis. The flank will be divided into two equal treatment areas where one side will receive multipolar radiofrequency with varipulse technology treatment and the other side will not.
Arm/Group | Cryolipolysis Treatment & Cryolipolysis With Legacy
Number analyzed (Participants) | 10
Number analyzed (flanks) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 9
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: General Improvement in Skin Laxity of the Flank Area
Description: Independent reviewer to identify the six month post-treatment photograph of the flank area treated with multi-polar radiofrequency, pulsed electro-magnetic fields and vacuum suction using the Global Aesthetic Improvement Scale (GAIS) where 3 = very much improved, 2 = much improved, 1 = improved, 0 = no change, -1 = worse, -2 = Much worse and -3 = very much worse.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: flank
Groups:
- Cryolipolysis Treatment & Cryolipolysis With Legacy: Each patient is their own control and one side will have only a cryolypolysis (Coolsculpt) treatment
Arm/Group | Cryolipolysis Treatment & Cryolipolysis With Legacy
Number analyzed (Participants) | 10
Number analyzed (flank) | 20
units on a scale
  Reviewer Cryoliposis GAIS at 6 month follow-up | 1.1 (1.0)
  Reviewer Cryolipolysis & RF, PEMF & varipulse GAIS | 2.1 (1.0)
Statistical Analysis 1: Comparison: Cryolipolysis Treatment & Cryolipolysis With Legacy; The null hypothesis was that the addition of the multipolar radiofrequency with varipulse technology treatment to the cryolipolysis treatment would not show visual improvement; Test type: Superiority — A significant improvement in skin laxity reduction is defined as a mean average increase in grade of 1 as per the GAIS; p < 0.01, Wilcoxon (Mann-Whitney); Used Wilcoxon Matched-Pairs Signed-Ranks test

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 11 months and 1 day.
Groups:
- ONE DEVICE USED - CoolSculpt Flank Side: Each patient is their own control and one side will have only a cryolypolysis (Coolsculpt) treatment
- TWO DEVICES USED - CoolSculpt and Venus Legacy Flank Side: Each patient is their own control and one side will have only a cryolypolysis (Coolsculpt) treatment while the other side will have both a cryolypolysis treatment and an RF, PEMF and Varipulse (Venus Legacy) treatment
Arm/Group | ONE DEVICE USED - CoolSculpt Flank Side | TWO DEVICES USED - CoolSculpt and Venus Legacy Flank Side
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ONE DEVICE USED - CoolSculpt Flank Side (N=10) | TWO DEVICES USED - CoolSculpt and Venus Legacy Flank Side (N=10)
Modest heat sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Modest erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
modest edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a pilot study to evaluate the treatment combination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No